CLINICAL TRIAL: NCT07272421
Title: A Three-Arm Randomized Controlled Trial Comparing Online ACT, Recuperation, and ACT Plus Vocational Support for Clinical Burnout
Brief Title: Comparing ACT, Recuperation, and ACT Plus Vocational Support for Clinical Burnout
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-05666-01
Record Dates: First submitted 2025-11-17; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Burnout; Clinical Burnout; Exhaustion Disorder
Keywords: ACT; Online; Burnout; Return To Work; Recovery
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: This is a three-arm, parallel-group, randomized controlled superiority trial evaluating three distinct 10-week psychological interventions for adults with clinical burnout. Participants are randomized in a 1:1:1 allocation ratio to:
  1. online Acceptance and Commitment Therapy (ACT),
  2. an online recuperation-focused program, or
  3. online ACT combined with structured vocational support.
Masking Description: This trial uses an open-label design in which participants and therapists are not masked to treatment allocation due to the nature of the psychological interventions. No additional parties are masked. Outcome data are collected through self-report questionnaires and registry-based sick-leave records, which are not influenced by treatment visibility. Statistical analysts will work with pseudonymized datasets, but this is for data protection rather than formal blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: ACT (Experimental): A 10-week online ACT program focusing on psychological flexibility, value clarification, and exposure to behaviors that maintain exhaustion (e.g., avoidance, perfectionism, rigid rules). Participants complete weekly digital modules with therapist guidance via written feedback and three brief video sessions.
  Interventions: Behavioral: ACT
- Arm 2: Recuperation (Active Comparator): A 10-week online program emphasizing rest, recuperation, and healthy daily routines. Content includes psychoeducation, sleep hygiene, pacing, relaxation, and gentle physical activity, without ACT-specific components. Participants complete weekly modules with therapist support through written feedback and three brief video sessions.
  Interventions: Behavioral: Recuperation
- Arm 3: ACT + vocational support (Active Comparator): A 10-week online ACT program combined with three additional sessions focused on work-related barriers and return-to-work planning. Participants receive weekly ACT modules with therapist guidance, three standard video sessions, and three vocational sessions delivered by licensed psychologists to create a structured, individualized RTW plan.
  Interventions: Behavioral: ACT; Behavioral: Vocational support

INTERVENTIONS:
Behavioral: ACT — The ACT intervention targets psychological flexibility using value clarification, functional analysis of stress-maintaining behaviors, mindfulness exercises, and structured exposure to avoidance, perfectionism, and rigid behavioral patterns associated with clinical burnout. The treatment content emphasizes reconnecting with personal values, increasing engagement in meaningful activities, and reducing ineffective coping strategies, such as excessive rest, overcontrol, and avoidance of work-related or emotionally difficult situations.
  Arms: Arm 1: ACT; Arm 3: ACT + vocational support
Behavioral: Recuperation — The recuperation intervention emphasizes restoring balance through rest, energy management, and healthy daily routines. Core content includes psychoeducation about stress and recovery, sleep hygiene, relaxation and breathing exercises, pacing strategies, gentle physical activity, and establishing structured routines for variation and recuperation. The treatment focuses on supporting restorative habits and reducing overload without using exposure, values work, or other ACT-specific methods.
  Arms: Arm 2: Recuperation
Behavioral: Vocational support — The vocational support component provides structured guidance to identify work-related barriers, clarify functional limitations, and develop a realistic, individualized return-to-work (RTW) plan. Content includes mapping job demands, exploring feasible work adjustments, formulating stepwise RTW goals, and identifying supports needed from the employer. Sessions focus on helping the participant create a written RTW plan that can be shared with relevant stakeholders.
  Arms: Arm 3: ACT + vocational support

SUMMARY:
This study compares three different online psychological treatments for people with clinical burnout (stress-related exhaustion) who are on sick leave or have major difficulties coping at work or in daily life. Many patients with burnout receive broad, recuperation-focused interventions (rest, stress reduction, lifestyle changes), but there is still no clearly evidence-based treatment or agreed clinical model. It is also known that returning to work can be difficult, and there is a need for more structured support.

In this trial, 210 adults in Sweden with clinical burnout will be randomly assigned to one of three 10-week, internet-based treatments:

Online Acceptance and Commitment Therapy (ACT) A structured, values-based CBT approach that focuses on helping participants clarify what matters to them, relate differently to difficult thoughts and feelings, and gradually re-engage in meaningful activities despite exhaustion.

Online Recuperation-focused treatment An active comparison condition that emphasizes rest, recuperation, and healthy daily routines. It provides psychoeducation and practical tools for sleep, relaxation, physical activity, pacing, and balance in everyday life, but does not include ACT-specific methods such as exposure or values work.

Online ACT plus Vocational Support The same ACT program as in group 1, together with three additional sessions with a licensed psychologist focused on work. These sessions help the participant identify work-related barriers, plan a gradual return-to-work (RTW), and formulate a written RTW plan that can be shared with the employer and treating physician.

All three treatments are delivered via a secure digital platform. Participants work through weekly online modules, receive written feedback from a therapist, and have three video sessions during the 10-week period. Clinical psychology students in their final semester deliver the ACT and recuperation treatments, and licensed psychologists deliver the ACT + vocational support condition.

The study has two primary aims:

1. to test whether online ACT reduces self-rated burnout symptoms more than the recuperation-focused treatment at the end of treatment, and
2. to test whether adding structured vocational support to ACT reduces the total number of registered sick-leave days in the year after treatment, compared with ACT alone.

Key secondary outcomes include perceived stress, depression, anxiety, insomnia, everyday memory problems, quality of life, functional impairment, treatment response and remission, treatment credibility and satisfaction, and cost-effectiveness. Outcomes are measured before treatment, weekly during treatment (for selected measures), immediately after treatment, and at 6- and 12-month follow-ups. Sick-leave data are obtained from the Swedish Social Insurance Agency.

To be eligible, participants must be 18 years or older, have symptoms consistent with clinical burnout (including pronounced fatigue and reduced stress tolerance after prolonged psychosocial stress), be on at least 25% sick leave or have marked functional impairment due to these symptoms, have a stable occupation or study situation, and be able to read and write Swedish. People with very long sick leave (more than two years), severe psychiatric conditions (such as severe depression, bipolar disorder, untreated PTSD, or psychosis), current substance abuse, or active suicidal ideation will not be included.

Potential risks include temporary increases in distress, fatigue, or symptom awareness when working with emotions, behavior change, or work-related issues. Participants are monitored closely through weekly questionnaires and therapist contact. If risk for self-harm or serious deterioration is detected, a licensed psychologist will perform a risk assessment and, if needed, refer the participant to appropriate health care.

The hope is that this study will identify effective, scalable, and theory-based online treatments for clinical burnout and clarify whether adding structured vocational support improves long-term work outcomes.

DETAILED DESCRIPTION:
Clinical burnout (also referred to as stress-related exhaustion) is a common reason for long-term sick leave in Sweden. Although many patients receive psychological or rehabilitative support, there is currently no established evidence-based treatment for clinical burnout, and the theoretical models guiding clinical care vary widely. Two dominant approaches in current practice are (1) recuperation-focused interventions emphasizing rest, balance, and lifestyle change, and (2) cognitive-behavioral approaches that aim to modify patterns of behavior and internal experience. Return-to-work (RTW) support is also widely regarded as important, yet structured, scalable, and well-defined RTW models tailored for burnout remain scarce.

This randomized controlled trial evaluates three 10-week online treatments for adults with clinical burnout:

1. Online Acceptance and Commitment Therapy (ACT) ACT is a contextual behavioral approach that aims to increase psychological flexibility-defined as the capacity to act in accordance with one's values while remaining open to difficult internal experiences. The intervention uses value clarification, behavior change strategies, mindfulness exercises, and structured exposure to behaviors that maintain exhaustion (e.g., avoidance, perfectionism, rigid rules around rest and activity). The program frames burnout as a crisis of engagement driven by excessive "musts" and "shoulds," helping participants reconnect with personally meaningful activities.
2. Online Recuperation-Focused Treatment This comparator is an active, credible intervention resembling what many patients receive in Swedish primary care. It focuses on rest, variation, energy monitoring, sleep hygiene, pacing, relaxation exercises, and general stress management. The treatment is primarily supportive and non-directive, emphasizing recuperation rather than behavioral exposure or value-guided change.
3. Online ACT plus Vocational Support This condition combines the ACT program with three additional sessions conducted by licensed psychologists focusing on work-related functioning. These sessions guide participants in mapping barriers to work participation, identifying feasible adjustments, and creating a written long-term RTW plan that can be shared with employers and treating physicians. This component is intended to support coordinated and gradual work reintegration.

Study Rationale Existing interventions for clinical burnout are often broad, multimodal, and resource-intensive. They may rely heavily on rest-based strategies and physiologically oriented explanations that risk reinforcing avoidance and passivity. ACT offers a theoretically coherent alternative that emphasizes behavioral re-engagement, values-based action, and psychological flexibility, which may be particularly relevant in burnout characterized by disengagement and rigid coping patterns.

At the same time, many patients with burnout struggle to return to work, and early coordination between the individual, employer, and health care system is often lacking. Integrating structured vocational support into an ACT treatment may help translate behavioral gains into improved work functioning.

Study Design This is a three-arm, parallel-group, randomized controlled superiority trial with a 1:1:1 allocation ratio. A total of 210 participants will be recruited across Sweden and randomized to one of the three interventions. Treatments are delivered over 10 weeks via the secure digital platform BASS. Each treatment includes 10 self-guided online modules, therapist feedback via weekly written chat, and three scheduled video sessions. The ACT + Vocational arm includes three additional vocational sessions.

All assessments, consent procedures, and follow-ups are conducted online. Registry data on sick leave will be obtained from the Swedish Social Insurance Agency for the 12 months following treatment, allowing for objective evaluation of long-term functional recovery.

Assessments occur at baseline, weekly during treatment (selected measures), mid-treatment, post-treatment, and at 6- and 12-month follow-up.

Intervention Delivery and Therapist Training Therapists in the ACT and Recuperation conditions are clinical psychology students in their final semester who have completed training in CBT. Licensed psychologists with experience in rehabilitation deliver the ACT + Vocational condition. All therapists receive structured protocols, two days of training, and weekly supervision to ensure consistent delivery and fidelity across conditions.

Primary Objectives Symptom reduction Evaluate whether ACT produces greater improvements in self-rated burnout symptoms than a recuperation-focused treatment at post-treatment and at follow-up.

Return-to-work outcomes Determine whether adding structured vocational support to ACT reduces the number of registered net sick-leave days during the 12 months after treatment.

Secondary and Exploratory Objectives Secondary objectives include comparing treatments on perceived stress, depression, anxiety, insomnia, everyday memory problems, quality of life, functional impairment, treatment adherence, treatment response and remission, and adverse effects. Process outcomes (e.g., psychological flexibility, recuperation behaviors, RTW self-efficacy) will also be assessed to examine change processes.

Economic evaluations will estimate cost-effectiveness from healthcare and societal perspectives. A qualitative sub-study will explore participants' experiences of ACT and, to a smaller extent, the other treatment arms.

Statistical Overview Repeated self-report outcomes will be analyzed using linear mixed-effects models with fixed effects for group, time, and group × time interactions, and random effects for participants. Sick-leave outcomes will be analyzed using negative binomial or Poisson regression models. All primary analyses will follow the intention-to-treat principle. Sensitivity, adjusted, and missing-data analyses (including multiple imputation) are planned.

The study is powered to detect small-to-moderate between-group effects on symptom trajectories and medium-sized differences in sick leave.

Data Monitoring and Safety Given the low-risk, non-pharmacological nature of the interventions, no independent data monitoring committee is established. Participants are monitored weekly, including automated alerts for worsening symptoms. Emergent risk (e.g., suicidal ideation) triggers same-day assessment by a licensed psychologist.

Adverse events will be recorded systematically during and after treatment.

Expected Contributions This study directly compares two theoretically distinct treatment models for clinical burnout and evaluates whether structured vocational support enhances functional recovery. It is among the first trials to assess an integrated, scalable ACT-based model for clinical burnout delivered entirely online. Findings may help identify effective strategies for reducing symptoms, supporting return to work, and informing the development of future evidence-based guidelines for clinical burnout.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Self-reported or clinically verified symptoms consistent with clinical burnout (e.g., pronounced fatigue, cognitive difficulties, and reduced stress tolerance following prolonged psychosocial stress)
* Currently on ≥25% sick leave and experiencing significant functional impairment in work or daily life due to these symptoms
* Stable occupation or engagement (employment or studies)
* Ability to read and write Swedish
* Daily access to the internet

Exclusion Criteria:

* Sick leave > 2 years for the current episode
* Severe acute psychiatric conditions, including: severe depression, bipolar disorder, untreated PTSD, schizophrenia, or other psychotic disorders
* Current substance abuse
* Active suicidal ideation (as assessed during clinical evaluation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Burnout Symptom Severity | Baseline (Week 0); weekly assessments during treatment (Weeks 1-10); mid-treatment (Week 5); post-treatment (Week 10, primary endpoint); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  This is one of two co-primary outcomes. Burnout symptoms will be assessed using the Shirom-Melamed Burnout Measure-12 (SMBM-12), a 12-item self-report scale measuring the core components of burnout: emotional and physical exhaustion (items 1-6) and cognitive/mental exhaustion (items 7-12). Each item is rated from 1 (almost never) to 7 (almost always). Items are averaged to produce a total mean score ranging from 1 (lowest level of burnout) to 7 (highest level of burnout). Higher scores indicate more severe burnout symptoms. Only the total mean score will be used as the primary outcome.
  Unit of Measure: SMBM-12 mean total score (1-7)
Net Sick-Leave Days | From post-treatment (Week 10) to 12-month follow-up (Month 12 post-treatment)
  This is one of two co-primary outcomes. This outcome reflects the total number of registered sick-leave days during the 12-month period following treatment. Data will be obtained from the Swedish Social Insurance Agency. Part-time sick leave will be converted into net days (e.g., 50% sick leave = 0.5 net day). Higher values indicate worse functional outcome (i.e., more days of sick leave).
  Unit of Measure: Net sick-leave days (0 to no upper limit)

SECONDARY OUTCOMES:
Perceived Stress | Baseline (Week 0); weekly assessments during treatment (Weeks 1-10); mid-treatment (Week 5); post-treatment (Week 10, primary endpoint); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Perceived stress will be measured using the Perceived Stress Scale-10 (PSS-10), a 10-item self-report questionnaire assessing the degree to which situations in one's life are appraised as stressful. Items are rated on a 0-4 scale and summed to a total score ranging from 0 (lowest perceived stress) to 40 (highest perceived stress). Higher scores indicate greater perceived stress.
Anxiety Symptoms Severity | Baseline (Week 0); mid-treatment (Week 5); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Anxiety severity will be measured using the Generalized Anxiety Disorder-7 (GAD-7), a 7-item self-report questionnaire. Each item is rated from 0 (not at all) to 3 (nearly every day). Items are summed to produce a total score ranging from 0 (no anxiety) to 21 (severe anxiety). Higher scores indicate greater anxiety severity.
  Unit of Measure: GAD-7 total score (0-21)
Depressive symptoms severity | Baseline (Week 0); mid-treatment (Week 5); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Depressive Symptom Severity will be measured using the Patient Health Questionnaire-9 (PHQ-9), a 9-item self-report scale. Each item is rated from 0 (not at all) to 3 (nearly every day). Items are summed to produce a total score ranging from 0 (no depressive symptoms) to 27 (severe depressive symptoms). Higher scores indicate greater depressive symptom severity.
  Unit of Measure: PHQ-9 total score (0-27)
Insomnia severity | Baseline (Week 0); mid-treatment (Week 5); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Sleep disturbance will be measured using the Insomnia Severity Index (ISI), a 7-item self-report scale assessing the severity and impact of insomnia symptoms. Each item is rated on a 0-4 scale, with response options reflecting increasing severity (e.g., from "no problem" to "very severe problem"). Item scores are summed to produce a total score ranging from 0 (no insomnia) to 28 (severe insomnia). Higher scores indicate greater sleep disturbance.
  Unit of Measure: ISI total score (0-28)
Health-Related Quality of Life | Baseline (Week 0); mid-treatment (Week 5); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Health-related quality of life will be measured using the EQ-5D-5L, which assesses five domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on a 5-level scale from 1 (no problems) to 5 (extreme problems). Responses are converted into a single index value based on the Swedish value set, ranging from values below 0 (states worse than death) to 1 (full health). Higher values indicate better health-related quality of life.
  Unit of Measure: EQ-5D-5L index value
Overall Quality of Life | Baseline (Week 0); mid-treatment (Week 5); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Quality of life will be measured using the Brunnsviken Brief Quality of Life Inventory (BBQ), which includes six life domains, each represented by a pair of items assessing importance and satisfaction. For each domain, the satisfaction rating is multiplied by the corresponding importance rating, producing a domain score ranging from 0 to 16. The total BBQ score is the sum of all weighted domain scores and ranges from 0 (lowest quality of life) to 96 (highest quality of life). Higher scores indicate better overall quality of life.
  Unit of Measure: BBQ weighted total score (0-96)
Treatment Satisfaction | Post-treatment (Week 10)
  Treatment satisfaction will be measured using the Client Satisfaction Questionnaire-8 (CSQ-8), an 8-item self-report scale assessing satisfaction with received treatment. Each item is rated from 1 to 4, with response anchors varying by item; however, in all items 1 reflects low satisfaction and 4 reflects high satisfaction. Item scores are summed to produce a total score ranging from 8 (lowest satisfaction) to 32 (highest satisfaction). Higher scores indicate greater treatment satisfaction.
  Unit of Measure: CSQ-8 total score (8-32)
Negative effects of Treatment | Post-treatment (Week 10)
  Potential adverse or unwanted effects of treatment will be assessed using the Negative Effects Questionnaire-20 (NEQ-20), a 20-item self-report measure. The NEQ-20 consists of five subscales, each scored by summing the items within the domain:
  Symptoms: items 1, 2, 3, 4, 6, 7, 8, 10 Quality: items 15, 16, 17, 18, 19, 20 Dependency: item 14 Stigma: items 9, 11 Hopelessness: items 5, 12, 13 Subscale scores are summed to produce a total score, with higher scores indicating a greater number or severity of negative effects. Response formats vary by item (e.g., presence, severity, or attribution).
  Unit of Measure: NEQ-20 total and subscale scores (higher = more negative effects).
Healthcare Utilization and Costs | Baseline (Week 0); mid-treatment (Week 5); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Healthcare utilization, productivity loss, and associated costs will be measured using the Trimbos and Institute of Medical Technology Cost Questionnaire for Psychiatry (TiC-P). The TiC-P assesses contacts with healthcare providers, medication use, informal care, and sickness absence/productivity loss. Cost categories will be calculated according to TiC-P scoring guidelines. Higher values reflect greater healthcare use or higher associated costs, depending on the component analyzed.
  Unit of Measure: TiC-P cost and utilization metrics

OTHER OUTCOMES:
Treatment Credibility and Expectancy | Week 1; mid-treatment (Week 5)
  Treatment credibility and outcome expectancy will be measured using the Credibility/Expectancy Questionnaire (CEQ), a 6-item self-report measure. Items 1-4 assess treatment credibility, and items 5-6 assess outcome expectancy. The CEQ uses two response formats (rating scales and percentage estimates), and subscale scores are calculated according to CEQ scoring guidelines. Higher scores indicate greater perceived credibility and expectancy.
  Unit of Measure: CEQ credibility and expectancy subscale scores (higher = greater credibility/expectancy)
Psychological Flexibility | Baseline (Week 0); weekly during treatment (Weeks 1-10); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Psychological flexibility will be assessed using the Psy-Flex scale, a 6-item self-report measure capturing core processes of psychological flexibility. Each item is rated from 1 (very inflexible) to 5 (very flexible). Items are summed to produce a total score ranging from 6 (lowest psychological flexibility) to 30 (highest psychological flexibility). Higher scores indicate greater psychological flexibility.
  Unit of Measure: Psy-Flex total score (6-30)
Recuperation Behaviors | Baseline (Week 0); weekly during treatment (Weeks 1-10); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Recuperation behaviors will be assessed using the Recuperation Behaviors Index (RPI-6), a formative process measure designed to capture multiple distinct aspects of recuperation. The index consists of six items representing complementary recuperation-related skills: detachment, relaxation, pacing, sleep protection, managing obligations, and prioritizing energy-restoring activities. Each item is rated from 1 (not at all true) to 7 (completely true), and items are summed to create a total score. Higher total scores indicate engagement in a broader set of recuperation behaviors.
  Content validity was established through expert ratings. The RPI-6 is included as a process measure to assess engagement in recuperation behaviors during treatment; full psychometric validation will be conducted in future research.
  Unit of Measure: RPI-6 total score
Return-to-Work Self-Efficacy | Baseline (Week 0); weekly during treatment (Weeks 1-10); post-treatment (Week 10); 6-month follow-up (Month 6 post-treatment); 12-month follow-up (Month 12 post-treatment)
  Description:
  Return-to-work self-efficacy will be assessed using a shortened version of the Self-Efficacy for Return to Work (SE-RTW) scale, originally developed by Lagerveld et al. (2010). The scale measures confidence in handling work demands, managing symptoms at work, and returning to or remaining in employment. Each item is rated on a 1-6 scale, from 1 = "strongly disagree" to 6 = "strongly agree." Items are summed to produce a total score, with higher scores indicating greater return-to-work self-efficacy.
  Unit of Measure: SE-RTW total score (higher = greater RTW self-efficacy)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data for all reported outcomes will be shared upon reasonable request after publication. Access will be granted to qualified researchers who provide a methodologically sound proposal and sign a data-sharing agreement. Data will be transferred through a secure repository in accordance with GDPR requirements.
Supporting Information: Study Protocol, SAP
Time Frame: Available beginning after publication of the primary results and for at least 5 years thereafter.
Access Criteria: Deidentified individual participant data and supporting documents will be accessible to qualified researchers affiliated with an academic institution or research organization. Access will be granted for purposes such as replication, meta-analysis, or other scientifically sound projects that align with the original study objectives.
  Researchers must submit a written request to the Principal Investigator describing the planned analyses and data requirements. Before access is granted, applicants must sign a data-sharing agreement ensuring compliance with ethical approvals, Swedish data protection legislation, and GDPR.
  Approved users will be able to access the data through a secure institutional repository at Uppsala University or via encrypted data transfer. Only deidentified datasets and approved supporting documents (e.g., protocol, analytic code) will be shared; no directly identifiable information will be provided.